CLINICAL TRIAL: NCT04439695
Title: A Phase 1, Observer-blinded, Randomized, Placebo-controlled, Parallel Group Study to Evaluate the Safety and Immunogenicity of KBP-V001 Quadrivalent Influenza Vaccine in Healthy Adults
Brief Title: Study to Evaluate the Safety and Immunogenicity of KBP-V001 Quadrivalent Influenza Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: KBio Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KBP-101
Record Dates: First submitted 2020-06-17; First posted 2020-06-19 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Influenza
Keywords: Influenza; Vaccine; Influenza Vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Contraceptives, Oral

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Low Dose KBP-V001 (Experimental): Subjects in this group will receive the low dose of KBP-V001.
  Interventions: Biological: Low dose
- Intermediate KBP-V001 (Experimental): Subjects in this group will receive the intermediate dose of KBP-V001.
  Interventions: Biological: Intermediate dose
- High Dose KBP-V001 (Experimental): Subjects in this group will receive the high dose of KBP-V001.
  Interventions: Biological: High dose
- Placebo (Placebo Comparator): Subjects in this group will receive placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Low dose — Low dose of KBP-V001
  Arms: Low Dose KBP-V001
Biological: Intermediate dose — Intermediate dose of KBP-V001
  Arms: Intermediate KBP-V001
Biological: High dose — High dose of KBP-V001
  Arms: High Dose KBP-V001
Biological: Placebo — Buffered Saline Solution
  Arms: Placebo

SUMMARY:
This is an observer-blinded, randomized, placebo-controlled, parallel group study to evaluate safety and immunogenicity of TAP-V001 quadrivalent influenza vaccine in healthy adult subjects.

DETAILED DESCRIPTION:
Subjects will be screened up to 14 days (Day -14 to Day 0) before randomization.

On the planned day of vaccination (Day 1), subjects will be randomized in a 1:1:1:1 ratio (N = 30 subjects/group) to receive study vaccine or placebo by intramuscular (IM) injection.

Approximately 5 subjects per group (N = 20) will be enrolled in parallel initially, and safety data through Day 8 will be collected. An Independent Data Monitoring Committee (IDMC) will convene to review Day 8 safety data before any additional subjects will be enrolled. If there are no safety concerns in the IDMC meeting, study enrollment will continue.

Blood and serum samples for safety laboratory tests and HAI titers will be obtained at baseline on Day 1 before administration of vaccine dose and after vaccination.

ELIGIBILITY:
Inclusion Criteria

1. Have read, understood, and signed the informed consent form (ICF)
2. Healthy adult males and females ages 18 to 49 years, inclusive at screening
3. Body mass index (BMI) of ≥18 and ≤34 kg/m2 at screening
4. Must be in general good health before study participation with no clinically relevant abnormalities that could interfere with study assessments
5. Women of childbearing potential (WOCBP) and men whose sexual partners are WOCBP must be able and willing to use at least 1 highly effective method of contraception during the study and for 3 months after the study completion. A female subject is considered to be a WOCBP after menarche and until she is in a postmenopausal state for 12 consecutive months (without an alternative medical cause) or otherwise permanently sterile (for which acceptable methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy).
6. Female subjects of childbearing potential must have a negative urine pregnancy test before vaccination
7. Must be able to attend all visits for the duration of the study and comply with all study procedures, including completion of Diary Card according to the study schedule.

Exclusion Criteria

1. History of an acute or chronic medical condition that, in the opinion of the investigator, would render vaccination unsafe or would interfere with the evaluation of responses.
2. History of ongoing clinical condition or medication or treatments that may adversely affect the immune system.
3. Individuals with any elevated (Grade 2 or higher) laboratory test assessed as clinically significant by investigator at screening
4. Individuals with any elevated (Grade 2 or higher) liver function enzyme at screening, regardless of the appraisal of clinical significance (cannot be retested to qualify for study). See below the criteria for excluding subjects with elevated liver enzymes:

   * Alanine aminotransferase (ALT)/aspartate aminotransferase (AST): >3 × upper limit of normal (ULN)
   * Total bilirubin: >2 × ULN
   * Alkaline phosphatase (ALP)/gamma-glutamyl transferase (GGT): >2.5 × ULN
5. Active neoplastic disease (excluding nonmelanoma skin cancer that was successfully treated) or a history of any hematological malignancy. For this criterion, "active" is defined as having received treatment within the past 5 years.
6. Long-term (greater than 2 weeks) use of oral or parenteral steroids or high-dose inhaled steroids (>800 μg/day of beclomethasone dipropionate or equivalent) within 6 months before screening (nasal and topical steroids are allowed)
7. History of autoimmune or inflammatory disease
8. Women currently pregnant, nursing, or planning a pregnancy between enrollment and 181 days after randomization
9. History of a previous serious adverse reaction to any influenza vaccine
10. History of Guillain-Barré Syndrome
11. History of anaphylactic-type reaction to injected vaccines
12. Known or suspected hypersensitivity to 1 or more of the components of TAP-V001
13. History of illicit drug use or alcohol abuse in the year before screening
14. Receipt of any influenza vaccine within 6 months before screening
15. Receipt of any vaccine within 1 month before screening
16. Acute illness or fever within 3 days before study enrollment (enrollment may be delayed for full recovery if acceptable to the investigator)
17. Individuals currently participating or planning to participate in a study that involves an experimental agent (vaccine, drug, biologic, device, or medication); or who have received an experimental agent within 1 month before enrollment in this study; or who expect to receive another experimental agent during participation in this study; or who intend to donate blood during the study period.
18. Receipt of immunoglobulin or another blood product within the 3 months before enrollment in this study or those who expect to receive immunoglobulin or another blood product during this study.
19. Individuals who plan to receive another vaccine, including seasonal influenza vaccine, during the entire 6-month study period.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2020-06-25 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-07-28 (Actual)

PRIMARY OUTCOMES:
Solicited administration site reactions | 7 days after vaccination
  Occurrences of Adverse Events
Solicited systemic events | 7 days after vaccination
  Occurrences of Adverse Events

SECONDARY OUTCOMES:
Number of Unsolicited Adverse Events | 43 days after vaccination
  Safety Endpoint
Number of Serious Adverse Events and Medically Attended Events | 181 days after vaccination
  Safety Endpoint
Vaccine HAI antibody Titers | Day 1, 29, 43, 181
  Vaccine HAI antibody Titers for each treatment group

CONTACTS AND LOCATIONS:
Overall Officials: Hugh Haydon, Study Director — Kentucky BioProcessing; Brandon Essink, MD, Principal Investigator — Meridian Clinical Research
Locations (1):
- Meridian Clinical Research, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No
Plan is to share study data by dosing group in publications